CLINICAL TRIAL: NCT02296775
Title: Comparative Pharmacokinetic, Pharmacodynamic, Safety and Efficacy Study of Three Anti-CD20 Monoclonal Antibodies in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RI-01-003
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Rituximab; Pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DRL_RI (Experimental)
  Interventions: Biological: DRL_RI
- Rituxan (Active Comparator)
  Interventions: Biological: Rituxan
- MabThera (Active Comparator)
  Interventions: Biological: MabThera

INTERVENTIONS:
Biological: DRL_RI — Two 1000 mg intravenous infusions, one each on Day 1 and Day 15
  Arms: DRL_RI
Biological: Rituxan — Two 1000 mg intravenous infusions, one each on Day 1 and Day 15
  Other Names: Rituximab
  Arms: Rituxan
Biological: MabThera — Two 1000 mg intravenous infusions, one each on Day 1 and Day 15
  Other Names: Rituximab
  Arms: MabThera

SUMMARY:
This study will compare the plasma pharmacokinetic profile and the change in disease activity score in patients with active rheumatoid arthritis following treatment with two 1000 mg doses of DRL_RI or one of two sources of rituximab (Rituxan® or MabThera®). Patients will also be monitored for safety, B cell depletion and recovery, and for the development of immune responses to the administered study drugs

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 18 to 65 years of age
2. Diagnosis of RA, according to ACR criteria (1987), of at least 6 months duration
3. At randomization, tender joint count ≥ 6 and swollen joint count ≥ 6
4. Evidence of at least moderate disease activity
5. Patients receiving oral or parenteral MTX with a dose of 15 to 25 mg per week when given alone or 10 to 25 mg per week in combination with additional non-biologic DMARD(s) for at least 6 months and on stable dose for at least 3 months
6. Patients must be on a stable dose of folic acid or equivalent (≥5 mg per week)
7. Chest X-ray not suggestive of any lung infections including pulmonary tuberculosis (TB)
8. Contraception required per protocol

Exclusion Criteria:

1. Prior therapy with

   * Rituximab, abatacept, tocilizumab, anakinra or an agent/antibody targeting CD20, CD19 or B cells
   * Tumor necrosis factor (TNF) alfa antagonists or other biologic DMARDs

   Other prior or concurrent therapies may also be excluded
2. Any clinically relevant abnormality detected on screening history, physical examination, clinical laboratory, chest X-ray, or electrocardiogram (ECG), other than values consistent with RA
3. Evidence of active, suspected or inadequately treated TB
4. Positive serological test for hepatitis C virus antibodies, hepatitis B surface antigen, hepatitis B core antibody, or human immunodeficiency virus
5. History of cardiovascular disease, history of stroke, or uncontrolled hypertension
6. History of lymphoproliferative disease or organ allograft
7. History of cancer (except for in situ cancer, excised, or limited stage, curatively treated cancer with no sign of disease for >5 years)
8. History of allergy (medication history) to any of the compounds used in the study
9. Pregnant or lactating women or women planning to become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- India (21):
  - Gurunank Care Hospital, Hyderabad, Andhra Pradesh
  - Care Hospitals, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences Ltd., Secunderabad, Andhra Pradesh
  - Yashoda Hospital, Secunderabad, Andhra Predesh
  - Shalby Hospitals, Ahmedabad, Gujarat
  - Government Medical College & New Civil Hospital, Surat, Gujarat
  - Chanre Rheumatology & Immunology Center & Research, Bangalore, Karnataka
  - Sushruta Multispeciality Hospital & Research Centre Pvt. Ltd, Hubli, Karnataka
  - Jagadguru Sri Shivarathreeshwara Hospital, Mysore, Karnataka
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute, Mumbai, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Deennath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Oyster & Pearl Hospital, Pune, Maharashtra
  - lnamdar Multispeciality Hospital, Pune, Maharashtra
  - Maulana Azad Medical College & Associated Lok Nayak Hospitals, New Delhi, National Capital Territory of Delhi
  - lndraprastha Apollo Hospitals, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College & Hosptial, Ludhiana, Punjab
  - S. R. Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Shri Nidaan Hospital & Hope Fertility Centre, Jaipur, Rajasthan
  - Apollo Specialty Hosptials, Madurai, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
- Ukraine (7):
  - Communal Healthcare Institution Kharkiv City Clinical Hospital #8, Kharkiv
  - State Institution National Scientific Center Acad. Strazhesko Institute of Cardiology of National Academy of Medical Science, Kyiv
  - State Institution D.F. Chebotariov Institute of Gerontology of NAMS of Ukraine, Kyiv
  - M.V. Sklifosovskyi Poltava Regional Clinical Hospital, Poltava
  - Vinnytsia M.I. Pyrogov Regional Clinical Hospital, Vinnytsia
  - Medical Clinical Investigational Center MC LLC Health Clinic, Vinnytsia
  - Communal Institution Zaporzhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia

REFERENCES:
- [Derived] Haridas VM, Katta R, Nalawade A, Kharkar S, Zhdan V, Garmish O, Lopez-Lazaro L, Batra SS, Kankanwadi S. Pharmacokinetic Similarity and Comparative Pharmacodynamics, Safety, Efficacy, and Immunogenicity of DRL_RI Versus Reference Rituximab in Biologics-Naive Patients with Moderate-to-Severe Rheumatoid Arthritis: A Double-Blind, Randomized, Three-Arm Study. BioDrugs. 2020 Apr;34(2):183-196. doi: 10.1007/s40259-020-00406-1. PMID 32052313

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 2 parts, a treatment and evaluation period (Part 1) and a recovery and follow-up period (Part 2).
  Study period was between November 2014 to June 2017 in a total of 29 sites across India and Ukraine.
Pre-assignment Details: The study was having 6 weeks screening period to accommodate 4 weeks washout/run-in stabilization and screening procedures.
Groups:
- DRL_RI (DRL Rituximab-Test Product Arm): DRL_RI 500 mg/50 mL solution in a single-use vial.
  On Day 1, all randomized patients were received one dose of 1000 mg of assigned study drug as a slow IV infusion. The second infusion was administered on Day 15.
- Rituxan® (US Licensed Reference Product): Rituxan® 500 mg/50 mL solution in a single-use vial. On Day 1, all randomized patients were received one dose of 1000 mg of assigned study drug as a slow IV infusion. The second infusion was administered on Day 15.
- MabThera® (EU Approved Reference Medicinal Product): MabThera® 500 mg/50 mL solution in a single-use vial.
  On Day 1, all randomized patients were received one dose of 1000 mg of assigned study drug as a slow IV infusion. The second infusion was administered on Day 15.
Period: Treatment and Evaluation
Arm/Group | DRL_RI (DRL Rituximab-Test Product Arm) | Rituxan® (US Licensed Reference Product) | MabThera® (EU Approved Reference Medicinal Product)
Started | 91 | 92 | 93
Completed | 87 | 84 | 83
Not Completed | 4 | 8 | 10
Period: Recovery and Follow-up
Arm/Group | DRL_RI (DRL Rituximab-Test Product Arm) | Rituxan® (US Licensed Reference Product) | MabThera® (EU Approved Reference Medicinal Product)
Started | 87 | 84 | 83
Completed | 82 | 79 | 79
Not Completed | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- DRL- Rituximab-DRL_RI; Rituxan® (US Licensed Reference Product): RP; MabThera® (EU Approved Reference Medicinal Product): RMP: On successful completion of the screening period, patients were randomized to 1 of the 3 treatment arms (DRL_RI, Rituxan®, or MabThera®) and administered 1000 mg of the study drug, one each on Day 1 and Day 15, while continuing their individual background stabilized DMARD regimen.
- Total: Total of all reporting groups
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP | Total
Number analyzed (Participants) | 91 | 92 | 93 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 92 | 93 | 276
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (10.96) | 44.0 (10.36) | 45.5 (10.41) | 44.5 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 81 | 81 | 243
  Male | 10 | 11 | 12 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Ukraine | 13 | 14 | 15 | 42
  India | 78 | 78 | 78 | 234
Disease Activity Score-C Reactive Protein (DAS28-CRP) [Mean (Standard Deviation); unit: Score on a scale] — Disease Activity Score (DAS) is used to assess improvement in disease activity in RA patients over time. The disease activity is interpreted as low (DAS <2.6), mild (2.6 to <3.2), moderate (3.2 to <5.1), and severe with DAS > 5.1. A DAS score between 0 and 2.6 corresponds to remission. The analysis of DAS28-CRP was based on a generalized estimating equation model in RA patients with DAS28 score > 3.2. Population: All patients who receive at least one dose of study drug and provide at least the baseline (pre-infusion of infusion and one post-baseline assessment of PD endpoints will be included in the PD population. Patients with relevant protocol deviations thought to affect the evaluations of PD endpoints will not be included in the PD population.
  Score on a scale
    number analyzed (Participants) | 86 | 86 | 85 | 257
    (all) | 6.031 (0.6702) | 5.719 (0.7603) | 5.831 (0.7024) | 5.786 (0.7233)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to 336 Hours (AUC0-336) Post First Dose
Description: PK samples were collected pre-infusion; 3 hours post infusion; EOI; and at 1, 6, 24, 48, 168 hours post End of Infusion. A PK sample at 336 hours post EOI were also to be collected after the second dose.
Time Frame: 2 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=218
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/ml
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 74 | 72 | 72
ug*h/ml | 49000 (27.1) | 49000 (25.4) | 51400 (24.1)

2. Primary Outcome: AUC0-∞ Over the Entire Course of Therapy (2 Doses) From Day 1 Through Week 16.
Description: as for outcome 1
Time Frame: 16 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=212
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/ml
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 73 | 71 | 68
ug*h/ml | 189000 (33.2) | 189000 (34.0) | 201000 (30.1)

3. Primary Outcome: Area Under Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t) (Second Dose).
Description: as for outcome 1
Time Frame: 16 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=220
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug*h/ml
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 76 | 71 | 73
ug*h/ml | 139000 (37.3) | 137000 (37.2) | 146000 (33.5)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) After First Dose
Description: Plasma concentration was measured at 0, 3, 4.25 (End of infusion (EOI)) ,1 (post- EOI), 6 (post-EOI) , 24 (post-EOI) , 48 (post-EOI) ,and 168 hours (post-EOI).
Time Frame: 2 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=218.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 74 | 72 | 72
ug/ml | 405.452 (24.5) | 388.017 (24.4) | 405.200 (30.1)

5. Secondary Outcome: Maximum Plasma Concentration (Cmax) After Second Dose
Description: Plasma concentration was measured at 0, 3, 4.25 (End of infusion (EOI)) ,1 (post- EOI),6 (post-EOI) , 24 (post-EOI) , 48 (post-EOI) , 168 (post-EOI), and 336 hours post EOI.
Time Frame: 2 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=224
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 78 | 72 | 74
ug/ml | 490.182 (28.1) | 470.237 (26.8) | 478.149 (24.7)

6. Secondary Outcome: Time to Cmax (Tmax) After First Dose.
Description: Plasma concentration was measured at 0, 3, 4.25 (End of infusion (EOI)) ,1 (post- EOI), 6 (post-EOI) , 24 (post-EOI) , 48 (post-EOI) , and 168 hours (post-EOI).
Time Frame: 2 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=218
Measure: Median (Full Range); unit: Hours
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 74 | 72 | 72
Hours | 5.25 [3.00 to 10.25] | 5.25 [4.25 to 10.33] | 5.25 [3.00 to 29.05]

7. Secondary Outcome: Time to Cmax (Tmax) After Second Dose
Description: as for outcome 6
Time Frame: 2 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=224
Measure: Median (Full Range); unit: Hours
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 78 | 72 | 74
Hours | 5.25 [3.00 to 10.33] | 5.25 [3.08 to 52.00] | 5.25 [3.00 to 27.25]

8. Secondary Outcome: Volume of Distribution (Vz)
Description: Plasma concentration was measured at 0, 3, 4.25 (End of infusion (EOI)) ,1 (post- EOI), 6 (post-EOI) , 24 (post-EOI) , 48 (post-EOI) , 168 (post-EOI), 336 hours (post-EOI), 4 weeks, 6 weeks, 8 weeks, 10 weeks, 14 weeks, 18 weeks, and 22 weeks relative to infusion.
Time Frame: 24 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=230
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 79 | 73 | 78
L | 5.69 (26.3) | 5.76 (23.1) | 5.55 (26.4)

9. Secondary Outcome: Systemic Clearance (CL)
Description: as for outcome 8
Time Frame: 24 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=230
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 79 | 73 | 78
L/day | 0.254 (33.2) | 0.254 (33.9) | 0.238 (30.0)

10. Secondary Outcome: Terminal Half-life (t1/2)
Description: as for outcome 8
Time Frame: 24 weeks
Population: Population numbers exclude ADA positive individuals and the total number analyzed is updated to n=230
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 79 | 73 | 78
h | 374 (30.1) | 378 (25.0) | 391 (23.9)

11. Secondary Outcome: Mean Change in Disease Activity Score-C Reactive Protein (DAS28-CRP) From Baseline Per Unit Time at Weeks 4
Description: In clinical studies, Disease Activity Score (DAS) is used to assess improvement in disease activity in RA patients over time. The assessment involved an examination of 28 joints for swelling, tenderness, blood C-reactive protein (CRP), and a one on one consultation between the patient and healthcare professional. The results were combined to produce a score which indicated how active the RA was at that particular time. The disease activity is interpreted as low (DAS <2.6), mild (2.6 to <3.2), moderate (3.2 to <5.1), and severe with DAS > 5.1. A DAS score between 0 and 2.6 corresponds to remission. The analysis of DAS28-CRP was based on a generalized estimating equation model in RA patients with DAS28 score > 3.2. The mean change was calculated from two time points (Value at 4 weeks minus baseline value).
Time Frame: Baseline and 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 85 | 85 | 83
units on a scale | -1.004 (0.9955) | -0.871 (0.7918) | -0.96 (0.9125)

12. Secondary Outcome: Mean Change in DAS28-CRP From Baseline Per Unit Time at 8 Weeks.
Description: In clinical studies, Disease Activity Score (DAS) is used to assess improvement in disease activity in RA patients over time. The assessment involved an examination of 28 joints for swelling, tenderness, blood C-reactive protein (CRP), and a one on one consultation between the patient and healthcare professional. The results were combined to produce a score which indicated how active the RA was at that particular time. The disease activity is interpreted as low (DAS <2.6), mild (2.6 to <3.2), moderate (3.2 to <5.1), and severe with DAS > 5.1. A DAS score between 0 and 2.6 corresponds to remission. The analysis of DAS28-CRP was based on a generalized estimating equation model in RA patients with DAS28 score > 3.2. The mean change was calculated from two time points (Value at 8 weeks minus baseline value).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 85 | 85 | 83
units on a scale | -1.379 (1.0274) | -1.192 (0.8635) | -1.424 (1.1764)

13. Secondary Outcome: Mean Change in DAS28-CRP From Baseline Per Unit Time at Week 12.
Description: In clinical studies, Disease Activity Score (DAS) is used to assess improvement in disease activity in RA patients over time. The assessment involved an examination of 28 joints for swelling, tenderness, blood C-reactive protein (CRP), and a one on one consultation between the patient and healthcare professional. The results were combined to produce a score which indicated how active the RA was at that particular time. The disease activity is interpreted as low (DAS <2.6), mild (2.6 to <3.2), moderate (3.2 to <5.1), and severe with DAS > 5.1. A DAS score between 0 and 2.6 corresponds to remission. The analysis of DAS28-CRP was based on a generalized estimating equation model in RA patients with DAS28 score > 3.2. The mean change was calculated from two time points (Value at 12 weeks minus baseline value).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 82 | 84 | 82
units on a scale | -1.652 (1.1405) | 1.443 (0.9648) | -1.718 (1.153)

14. Secondary Outcome: Mean Change in Disease Activity Score- C Reactive Protein (DAS28-CRP) From Baseline Per Unit Time at Week 16.
Description: In clinical studies, Disease Activity Score (DAS) is used to assess improvement in disease activity in RA patients over time. The assessment involved an examination of 28 joints for swelling, tenderness, blood C-reactive protein (CRP), and a one on one consultation between the patient and healthcare professional. The results were combined to produce a score which indicated how active the RA was at that particular time. The disease activity is interpreted as low (DAS <2.6), mild (2.6 to <3.2), moderate (3.2 to <5.1), and severe with DAS > 5.1. A DAS score between 0 and 2.6 corresponds to remission. The analysis of DAS28-CRP was based on a generalized estimating equation model in RA patients with DAS28 score > 3.2. The mean change was calculated from two time points (Value at 16 weeks minus baseline value).
Time Frame: Baseline and 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 83 | 85 | 82
units on a scale | -1.892 (1.1257) | -1.49 (1.0222) | -1.814 (1.2105)

15. Secondary Outcome: Percentage of Patients With B-cell Counts 20% Below the Lower Limit of Normal
Description: The time to depletion and repletion of peripheral blood cell counts (determined by CD19+ cell counts) as well as the B-cell counts at selected time points (taking into consideration the patient baseline count) were used to assess the PD of the study drugs.
Time Frame: 48 hours
Measure: Number; unit: Percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 86 | 87 | 86
Percentage of participants | 98.8 | 100 | 100

16. Secondary Outcome: Percentage of Patients With Peripheral B-cell Counts Depletion at Week 16.
Description: Analysis of the PD parameter peripheral B-Cell count was performed by evaluating the 95% CI for the difference between treatment arms in the percentage of patients with B-cell depletion at 48 hours after dose 1, Week 16, and at Week 24. Percentage of patients with B-cell repletion at each evaluation time is also reported and descriptively compared.
Time Frame: 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 86 | 87 | 86
percentage of participants | 10.0 | 4.9 | 10.1

17. Secondary Outcome: Percentage of Patients With Peripheral B-cell Counts Depletion at Week 24.
Description: as for outcome 16
Time Frame: 24 weeks
Measure: Number; unit: percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 86 | 87 | 86
percentage of participants | 0.0 | 3.7 | 1.3

18. Secondary Outcome: Percentage of Patients With ACR20 at Week 24
Description: Percentage of the patients with at least 20% improvement in counts of tender, swollen joints and in 3 of the following: patient's assessment of pain, patient's global assessment of disease activity, patient's assessment of physical function, the physician's global assessment of disease activity, and acute phase reactant. Adjusted response rates for the treatment arms using the logistic regression analysis including treatment, gender and region as fixed effects and patients as random effect in the model.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 59 | 56 | 54
Percentage of participants | 72 | 69.1 | 68.4

19. Secondary Outcome: Percentage of Patients With ACR50 at Week 24
Description: Percentage of the patients with at least 50% improvement in counts of tender, swollen joints and in 3 of the following: patient's assessment of pain, patient's global assessment of disease activity, patient's assessment of physical function, the physician's global assessment of disease activity, and acute phase reactant. Adjusted Response rates for the treatment arms using the logistic regression analysis including treatment, gender and region as fixed effects and patients as random effect in the model.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 36 | 32 | 34
Percentage of participants | 43.9 | 39.5 | 43.0

20. Secondary Outcome: Percentage of Patients With ACR70 Response at Week 24
Description: Percentage of the patients with at least 70% improvement in counts of tender, swollen joints and in 3 of the following: patient's assessment of pain, patient's global assessment of disease activity, patient's assessment of physical function, the physician's global assessment of disease activity, and acute phase reactant. Adjusted Response rates for the treatment arms using the logistic regression analysis including treatment, gender and region as fixed effects and patients as random effect in the model.
Time Frame: 24 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 14 | 12 | 12
Percentage of participants | 17.1 | 14.8 | 15.2

21. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24.
Description: The health assessment questionnaire disability index (HAQ-DI) was assessed at Week 24. The disability assessment component of the HAQ, the HAQ-DI, assessed a patient's level of functional ability and included questions about fine movements of the upper extremities, locomotor activities of the lower extremities, and activities that involved both upper and lower extremities. There were 20 questions in 8 categories of functioning which represented a comprehensive set of functional activities-dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The stem of each item asked over the past week "Were you able to" perform a particular task. The patient's responses were made on a scale from 0 (no disability) to 3 (completely disabled). Each category contained at least 2 specific component questions.
  Physical function was measured using the HAQ-DI Scores, which range from 0-3, with lower scores reflecting better physical function and thus, less disability.
Time Frame: 24 weeks
Measure: Geometric Mean (Standard Deviation); unit: score on a scale
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
Number analyzed (Participants) | 82 | 81 | 79
score on a scale | 0.742 (0.60603) | 0.691 (0.62598) | 0.726 (0.5659)

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (52 weeks)
Arm/Group | DRL- Rituximab-DRL_RI | Rituxan® (US Licensed Reference Product): RP | MabThera® (EU Approved Reference Medicinal Product): RMP
All-Cause Mortality (participants affected / at risk) | 2/91 | 0/92 | 0/93
Serious Adverse Events (participants affected / at risk) | 3/91 | 5/92 | 10/93
Other Adverse Events (participants affected / at risk) | 60/91 | 58/92 | 66/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRL- Rituximab-DRL_RI (N=91) | Rituxan® (US Licensed Reference Product): RP (N=92) | MabThera® (EU Approved Reference Medicinal Product): RMP (N=93)
H1N1 Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Penumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Febile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRL- Rituximab-DRL_RI (N=91) | Rituxan® (US Licensed Reference Product): RP (N=92) | MabThera® (EU Approved Reference Medicinal Product): RMP (N=93)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 3 (3) | 5 (5) — All AE's are listed as TEAE's for this study
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (5) | 1 (1) — All AE's are listed as TEAE's for this study
Urinary Tract Infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2) — All AE's are listed as TEAE's for this study
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) — All AE's are listed as TEAE's for this study
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — All AE's are listed as TEAE's for this study
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Hyperchlorhydia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) — All AE's are listed as TEAE's for this study
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) — All AE's are listed as TEAE's for this study
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) — All AE's are listed as TEAE's for this study
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Blood creatnine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 2 (2) — All AE's are listed as TEAE's for this study
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) — All AE's are listed as TEAE's for this study
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Pyrexia (General disorders) | 2 (2) | 4 (4) | 3 (3) — All AE's are listed as TEAE's for this study
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Generalized oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) — All AE's are listed as TEAE's for this study
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) — All AE's are listed as TEAE's for this study
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 3 (3) — All AE's are listed as TEAE's for this study
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (2) — All AE's are listed as TEAE's for this study
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) — All AE's are listed as TEAE's for this study
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — All AE's are listed as TEAE's for this study
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study.
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) | 1 (1) — All AEs are listed as TEAEs for this study
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) — All AEs are listed as TEAEs for this study
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) — All AEs are listed as TEAEs for this study
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) — All AEs are listed as TEAEs for this study
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — All AEs are listed as TEAEs for this study.
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1) — All AEs are listed as TEAEs for this study
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) — All AEs are listed as TEAEs for this study
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — All AEs are listed as TEAEs for this study
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) — All AEs are listed as TEAEs for this study
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — All AEs are listed as TEAEs for this study
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — All AEs are listed as TEAEs for this study
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) — All AEs are listed as TEAEs for this study
Cervicobrachial syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) — All AEs are listed as TEAEs for this study
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Trachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) — All AEs are listed as TEAEs for this study
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) — All AEs are listed as TEAEs for this study
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — All AEs are listed as TEAEs for this study
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — All AEs are listed as TEAEs for this study
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — All AEs are listed as TEAEs for this study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes